CLINICAL TRIAL: NCT02658110
Title: Acute Metabolic and Appetite Responses to Altered Timing of Whey Protein Ingestion in Overweight and Obese Males
Brief Title: Metabolic and Appetite Responses to Altered Timing of Whey Protein Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HLSDA020415
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Obesity, Abdominal
Keywords: Postprandial glycemia; Metabolic health measures
MeSH Terms: conditions — Obesity, Abdominal | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Non Protein Trial (Sham Comparator): Mixed Macronutrient Breakfast Meal and Mixed Macronutrient Lunch Meal served without additional whey protein
  Interventions: Other: Mixed Macronutrient Breakfast Meal; Other: Mixed Macronutrient Lunch Meal
- Preload Trial (Experimental): Whey protein (20g) administered 15 minutes prior to Mixed Macronutrient Breakfast Meal
  Interventions: Dietary Supplement: Whey Protein; Other: Mixed Macronutrient Breakfast Meal; Other: Mixed Macronutrient Lunch Meal
- With Meal Trial (Experimental): Whey protein (20g) administered alongside Mixed Macronutrient Breakfast Meal
  Interventions: Dietary Supplement: Whey Protein; Other: Mixed Macronutrient Breakfast Meal; Other: Mixed Macronutrient Lunch Meal
- Post Meal Trial (Experimental): Whey protein (20g) administered 15 minutes after Mixed Macronutrient Breakfast Meal
  Interventions: Dietary Supplement: Whey Protein; Other: Mixed Macronutrient Breakfast Meal; Other: Mixed Macronutrient Lunch Meal

INTERVENTIONS:
Dietary Supplement: Whey Protein — 20 g whey protein isolate (Arla Foods Ingredients Group) added to 200ml water and served as a beverage
  Arms: Post Meal Trial; Preload Trial; With Meal Trial
Other: Mixed Macronutrient Breakfast Meal — A standardised mixed-macronutrient breakfast served to all participants. The macronutrient distribution of the breakfast is 13% protein, 70% carbohydrate, 17% fat (1958 kJ; 468 kcal total)
Other: Mixed Macronutrient Lunch Meal — A standardised mixed-macronutrient lunch served to all participants. The macronutrient distribution of the lunch is 14% protein, 51% carbohydrate, 35% fat (3506 kJ; 838 kcal total)

SUMMARY:
The proposed study aims to determine the metabolic and appetite responses to standard breakfast and lunch meals whilst altering the timing of whey protein supplementation. Currently, the designs implemented in many studies mean that it is unclear whether an optimum time for whey protein consumption exists in order to promote the greatest acute health benefits. A number of studies have investigated the effects of whey protein when consumed as a preload to a subsequent meal, whilst benefits have also been shown when whey protein is ingested with a meal. The proposed study will therefore investigate strategies of whey protein supplementation that vary in their practical applicability, using meals that reflect regular eating behaviours throughout the population in a sample of overweight/obese individuals.

Findings from this study may provide important information regarding the efficacy of whey protein supplementation before, during and after a composite meal, and its effect on the handling of a subsequent mixed-macronutrient meal.

DETAILED DESCRIPTION:
A randomised crossover design shall be implemented, whereby all participants complete 4 trials separated by a minimum of 3 days. On all visits participants shall consume a standardised mixed-macronutrient breakfast meal, followed 180 minutes later by consumption of a standard lunch meal. The timing of additional protein supplementation shall vary by trial, with participants consuming a shake containing 20g whey protein isolate either as a preload (15 minutes prior to breakfast), alongside the breakfast meal, or 15 minutes following breakfast consumption. A control trial shall also be completed without additional protein supplementation. At all supplementation time points participants shall consume either a flavoured whey protein shake or a flavoured water isovolumetric beverage ensuring that they remain blinded to the condition. Venous and capillary blood samples and visual analogue scales (for determination of subjective appetite sensations) shall be taken at regular intervals following both meals while the participant is rested.

ELIGIBILITY:
Criteria for inclusion are as follows:

* Male
* Aged 18-55 years
* Abdominal obesity (Waist circumference > 102 cm)
* Sedentary (not currently participating in structured physical activity)

Criteria for exclusion are as follows:

* Metabolic disease or current illness
* Regular breakfast skipper
* Food allergies/intolerances
* Eating disorders
* Smoking

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose responses | 0-360 minutes post breakfast
  Blood glucose concentration determined in whole blood sampled at regular intervals post-breakfast and post-lunch

SECONDARY OUTCOMES:
Acute subjective appetite responses | 0-360 minutes post breakfast
  Subjective appetite ratings determined from Visual Analogue Scales sampled at regular intervals

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Study Director — Northumbria University
Locations (1):
- Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No